CLINICAL TRIAL: NCT05461482
Title: CLINTERVENTIONAL Trial: A Randomized Controlled Two-arm Trial to Evaluate the Impact of Clinical Consultations and Audiovisual Tools in Patients Who Are Going to Undergo Interventional Radiology Procedures.
Brief Title: CLINTERVENTIONAL Trial: Impact of Clinical Consultations and Audiovisual Tools in Interventional Radiology
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maimónides Biomedical Research Institute of Córdoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Analisis RVI
Record Dates: First submitted 2022-04-20; First posted 2022-07-18 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-10

CONDITIONS: Interventional Radiology; Physician-Patient Relations; Communication; Physician's Practice Patterns; Patient Satisfaction
MeSH Terms: conditions — Communication; Patient Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): The physician requesting the intervention will be responsible for informing the patient, explaining the purpose of the intervention, its risks and benefits, and possible alternatives and doubts related to the intervention.
- Experimental group (Experimental): In addition to the information provided by the referring physician, an interventional radiologist will assist the patient in a consultation before the intervention to inform him, explaining the objective of the intervention, its risks and benefits, and possible alternatives and doubts related to the intervention. In this group, educational videos will be used, one for each type of intervention, which will complement the explanations of the physician. The videos will aim to present in an understandable way the preparation for the intervention, its objective, the benefits and risks that derive from it and what you can expect once it has been carried out. Patients will have access to the videos before attending the consultation and will view them before being seen by the interventional radiologist.
  Interventions: Other: Pre-procedural consultation and audiovisual tools

INTERVENTIONS:
Other: Pre-procedural consultation and audiovisual tools — In addition to the information provided by the referring physician, an interventional radiologist will assist the patient in a consultation before the intervention to inform him, explaining the objective of the intervention, its risks and benefits, and possible alternatives and doubts related to the intervention. In this group, educational videos will be used, one for each type of intervention, which will complement the explanations of the physician. The videos will aim to present in an understandable way the preparation for the intervention, its objective, the benefits and risks that derive from it and what you can expect once it has been carried out. Patients will have access to the videos before attending the consultation and will view them before being seen by the interventional radiologist.
  Arms: Experimental group

SUMMARY:
* Objectives: To assess whether the implementation of pre-procedural consultations and the use of explanatory audiovisual tools prior to performing Vascular and Interventional Radiology procedures improve the understanding of interventions by patients, improve satisfaction with the information provided and reduce anxiety experienced by the procedure.
* Methods: We will conduct a two-arm randomized clinical trial that will include patients undergoing Vascular and Interventional Radiology procedures. After consent to participation by signing the informed consent, participants will be randomly assigned to the control group (patients to whom the information about the procedure is provided by the requesting physician) and to the experimental group (patients who, in addition to being informed by the requesting physicians, are attended by interventional radiologists in consultation after previously viewing explanatory videos of the interventions). Multi-choice questionnaires will be used to assess understanding and knowledge of the interventions and validated scales to measure satisfaction with the information provided and anxiety experienced. Knowledge and understanding of the intervention, satisfaction with the information transmitted and the method of transmission, as well as anxiety related to the intervention will be compared between the control group and the experimental group. The Student's t-test and the Mann-Whitney test will be used for the comparison of quantitative variables and the chi-square test and Fisher's exact test for the comparison of qualitative variables. Regression analysis will be used to evaluate associations between variables.
* Expected results: To demonstrate that the implementation of pre-procedural consultations attended by interventional radiologists and the use of educational audiovisual tools prior to performing Vascular and Interventional Radiology procedures improve the understanding of interventions by patients, their satisfaction with the information provided and reduces the anxiety experienced for the procedure.
* Potential impact: It is the first clinical trial that analyzes the usefulness of pre-procedural consultations and audiovisual tools in Vascular and Interventional Radiology, so its results will be very interesting to help standardize clinical practice in Vascular and Interventional Radiology.

ELIGIBILITY:
To be eligible, each patient must meet one of the inclusion criteria and none of the exclusion criteria.

Inclusion Criteria:

* Patients who are going to undergo one of the following elective vascular interventional procedures: tunneled cuffed catheter placement, fistulography and endovascular treatment of hemodialysis arteriovenous fistulas, vascular recanalization procedures and vascular embolization procedures.
* Patients undergoing one of the following elective nonvascular interventional procedures: image-guided percutaneous biopsies, percutaneous fluid and abscess drainage, percutaneous transhepatic biliary drainage and percutaneous nephrostomy.

Exclusion Criteria:

* Patients under 18 years of age.
* Patients who require the participation of a third party for informed consent.
* Pregnant patients.
* Patients undergoing urgent interventional procedures.
* Patients with allergy or intolerance to mepivacaine, tramadol, midazolam or fentanyl.
* Patients who do not understand and speak Spanish properly.
* Patients with deafness or blindness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 428 (Estimated)
Dates: Start 2022-08-31 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Change in Knowledge from baseline to immediately preoperatively using a multi-choice questionnaire. Where the patient's knowledge was assessed related to the intervention. | From baseline at preoperative assessment to immediately preoperatively: 24 hours.
  It will be assessed if the preparation for the intervention, the indication, the intervention itself, the subsequent care and the benefits, risks and alternatives are known and understood. It will be analyzed using a multi-choice questionnaire.
Change in Anxiety from baseline to immediately preoperatively using a Visual analogue scale (0-10) and State-Trait Anxiety Inventory (20-80). | From baseline at preoperative assessment to immediately preoperatively: 24 hours.
  It will be assessed if the preparation for the intervention, the indication, the intervention itself, the subsequent care and the benefits, risks and alternatives are known and understood. It will be analyzed using a multi-choice questionnaire.
Change in satisfaction from baseline to immediately preoperatively using a Visual analogue scale (0-10). | From baseline at preoperative assessment to immediately preoperatively: 24 hours.
  It will be assessed if the preparation for the intervention, the indication, the intervention itself, the subsequent care and the benefits, risks and alternatives are known and understood. It will be analyzed using a multi-choice questionnaire.

SECONDARY OUTCOMES:
Assessment the association between all of variables through a descriptive analysis using SPSS. | Through study completion: 18 months
  It will be assessed the association between demographic variables, type of intervention, personal history, intervention group, anxiety related to the intervention, level of knowledge and understanding of the intervention, type of anesthesia, and degree of sedation with the pain intensity during the intervention, with the level of tolerance of the intervention and with the level of satisfaction with the intervention performed
To contrast differences in the variables of both arms through a descriptive analysis using SPSS. | Through study completion: 18 months
  Comparative analysis of the duration of the intervention, the intensity of the pain perceived by the patient during the procedure, the level of tolerance of the intervention and the level of satisfaction with the intervention carried out in the two groups of patients.

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Blas García Jurado, MD, Principal Investigator — Reina Sofia University Hospital
Locations (1):
- Hospital Universitario Reina Sofia, Córdoba, Spain

REFERENCES:
- [Derived] Garcia Jurado PB, Espejo Herrero JJ, Lombardo Galera MS, Perez Montilla ME, Barranco Acosta S, Garcia-Revillo Garcia J, Font Ugalde P, Alvarez Benito M. Impact of the clinical role of interventional radiologists: results of the CLINTERVENTIONAL randomized controlled trial. Eur Radiol. 2025 Dec;35(12):7658-7668. doi: 10.1007/s00330-025-11757-0. Epub 2025 Jun 17. PMID 40526354
- [Derived] Garcia Jurado PB, Espejo Herrero JJ, Lombardo Galera MS, Perez Montilla ME, Barranco Acosta S, Garcia-Revillo J, Font Ugalde P, Alvarez Benito M. CLINTERVENTIONAL protocol: a randomized controlled trial to evaluate clinical consultations and audiovisual tools for interventional radiology. Eur Radiol Exp. 2025 Jan 15;9(1):6. doi: 10.1186/s41747-024-00545-y. PMID 39812733